CLINICAL TRIAL: NCT00920907
Title: A Randomized, Parallel, Open-Label Study to Compare the Pharmacokinetics of Ipilimumab (BMS-734016) Process C to Process B in Subjects With Advanced Melanoma
Brief Title: Comparison of Ipilimumab Manufactured by 2 Different Processes in Participants With Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Medarex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-087
Record Dates: First submitted 2009-06-09; First posted 2009-06-15 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ipilimumab (Process B) (Experimental): Reference
  Interventions: Biological: Ipilimumab
- Ipilimumab (Process C) (Experimental): Test
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab — Solution, Intravenous, 10 mg/kg, Every 3 weeks (up to 4 doses) in induction phase, every 12 weeks in maintenance phase, 48 weeks
  Other Names: BMS-734016; MDX010

SUMMARY:
The purpose of this clinical research study is to compare pharmacokinetics of ipilimumab manufactured by two different processes

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of malignant melanoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Measurable/evaluable disease per modified World Health Organization (mWHO) criteria

Exclusion Criteria:

* Active Brain Metastasis
* Primary ocular or mucosal melanoma
* Prior Autoimmune disease
* Inadequate hematologic, hepatic or renal function
* Use of immunosuppressants
* Prior treatment with a CD137 agonist or cytotoxic T lymphocyte antigen 4 (CTLA-4) inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - The Angeles Clinic & Research Inst., Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - St Luke'S Hospital And Health Network, Bethlehem, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Kitano S, Postow MA, Ziegler CG, Kuk D, Panageas KS, Cortez C, Rasalan T, Adamow M, Yuan J, Wong P, Altan-Bonnet G, Wolchok JD, Lesokhin AM. Computational algorithm-driven evaluation of monocytic myeloid-derived suppressor cell frequency for prediction of clinical outcomes. Cancer Immunol Res. 2014 Aug;2(8):812-21. doi: 10.1158/2326-6066.CIR-14-0013. Epub 2014 May 20. PMID 24844912
- [Derived] Iwama S, De Remigis A, Callahan MK, Slovin SF, Wolchok JD, Caturegli P. Pituitary expression of CTLA-4 mediates hypophysitis secondary to administration of CTLA-4 blocking antibody. Sci Transl Med. 2014 Apr 2;6(230):230ra45. doi: 10.1126/scitranslmed.3008002. PMID 24695685
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started August 3, 2009, ended October 31, 2012; Induction Phase (Weeks 1, 4, 7, 10), Maintenance Phase (participants without immune-related progressive disease (irPD) received ipilimumab every 12 weeks until disease progression, toxicity, pregnancy, death, withdrew consent, lost to follow up); Patients followed for 10 weeks post last dose.
Pre-assignment Details: 99 participants enrolled; 75 participants randomized and treated. 24 participants not treated due to violations of inclusion or exclusion criteria.
Groups:
- Ipilimumab (Process B): Intravenous (IV) solution of 10 milligrams (mg) ipilimumab per kilogram (kg) of body weight was given once every 3 weeks (up to 4 doses) in the induction phase (Weeks 1, 4, 7, and 10); it was given once every 12 weeks in the maintenance phase for 48 weeks. In Process B, ipilimumab was manufactured by the Lonza company using material from transfectoma cell line.
- Ipilimumab (Process C): Intravenous (IV) solution of 10 milligrams (mg)ipilimumab per kilogram (kg) of body weight was given once every 3 weeks (up to 4 doses) in the induction phase (Weeks 1, 4, 7, and 10); it was given once every 12 weeks in the maintenance phase for 48 weeks. In Process C, ipilimumab was manufactured by Sponsor using material from a sub-clone of the original transfectoma cell line, modified cell culture and purification steps.
Period: Induction Period
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Started | 37 | 38
Completed | 15 | 16
Not Completed | 22 | 22
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 1
Not completed — Disease Progression | 12 | 11
Not completed — Study Drug Toxicity | 8 | 6
Not completed — No longer meets study criteria | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Maintenance Period
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Started | 15 | 15 (1 patient completed Induction phase but discontinued the study prior to start of maintenance phase.)
Completed | 3 (All participants who entered Maintenance were treated with study drug.) | 2 (2 participants who entered Maintenance Period did not receive study drug during the period.)
Not Completed | 12 | 13
Not completed — Disease Progression | 3 | 7
Not completed — Administrative (study closure) | 7 | 2
Not completed — Study Drug Toxicity | 0 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ipilimumab (Process B): 10 mg/kg ipilimumab was given IV once every 3 weeks (up to 4 doses) in the induction phase (Weeks 1, 4, 7, and 10); it was given once every 12 weeks in the maintenance phase for 48 weeks. In Process B, ipilimumab was manufactured by Lonza using material from transfectoma cell line.
- Ipilimumab (Process C): 10 mg/kg ipilimumab was given IV once every 3 weeks (up to 4 doses) in the induction phase (Weeks 1, 4, 7, and 10); it was given once every 12 weeks in the maintenance phase for 48 weeks. In Process C, ipilimumab was manufactured by the Sponsor using material from a sub-clone of the original transfectoma cell line, modified cell culture and purification steps.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C) | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14) | 59 (12) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 25 | 24 | 49
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75
Body Weight [Mean (Standard Deviation); unit: kg] — Body weight measured in kilograms (kg).
  kg | 81.3 (13.4) | 80.7 (13.3) | 81.0 (13.3)
Eastern Cooperative Oncology Group (ECOG) [Number; unit: participants] — ECOG performance: 0= Fully active, able to carry on all pre-disease performance without restriction;1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or Chair; 5=Dead
  participants
    ECOG=0 | 25 | 21 | 46
    ECOG=1 | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Ipilimumab Manufactured by Process C Relative to the Cmax of Ipilimumab Manufactured by Process B - Evaluable Pharmacokinetic Population
Description: Single-dose Pharmacokinetic (PK) parameters of ipilimumab were derived from serum concentration versus time data. Cmax was measured from first dose to end of the induction period (4 doses) as micrograms per milliliter (μg/mL). Samples were obtained at 0 hour (predose) on Days 1, 2, 3, 4, and Weeks 2, 3, 4, 7, and 10; Day 1, samples were also obtained 1 h 30 minutes (min), 2 h, 2 h 30 min, 3 h 30 min, 4 h 30 min, and 6 h post dose. In calculating PK parameters, predose concentrations and concentrations prior to first quantifiable concentration below the lower limit of quantitation (LLOQ) were treated as "missing" for the calculation of summary statistics. Drug was quantitatively determined in serum by an enzyme-linked immunosorbent assay (ELISA). Individual PK parameter values were derived by non-compartmental methods using a validated PK analysis program (Kinetica™ 4.4.1 within eToolbox [version 2.6.1]).
Time Frame: Day 1 to Day 84
Population: Pharmacokinetic (PK) evaluable Population: All participants who received at least one dose of drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 36 | 38
μg/mL | 252.68 (29) | 251.26 (24)
Statistical Analysis 1: Comparison: Ipilimumab (Process B) vs Ipilimumab (Process C); Biocomparability of ipilimumab Process C to ipilimumab Process B was concluded if the 90% confidence intervals (CIs) for the ratio of geometric means for Cmax were contained within 80% to 125%; Test type: Superiority or Other; Least squared linear regression; Ratio of adjusted geometric mean = 1.010, 90% CI 2-sided [0.916 to 1.114]

2. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax) of Ipilimumab Manufactured by Process C Relative to the Tmax of Ipilimumab Manufactured by Process B - Evaluable Pharmacokinetic Population
Description: The single-dose Pharmacokinetic parameters of ipilimumab were derived from serum concentration versus time data. Tmax was measured from first dose to end of the induction period (4 doses) in hours (h). Samples were obtained at 0 h (predose) on Days 1, 2, 3, 4, and Weeks 2, 3, 4, 7, and 10; Day 1, samples were also obtained 1 h 30 minutes (min), 2 h, 2 h 30 min, 3 h 30 min, 4 h 30 min, and 6 h post dose. In calculating PK parameters, predose concentrations and concentrations prior to first quantifiable concentration below the lower limit of quantitation (LLOQ) were treated as "missing" for the calculation of summary statistics. Drug was quantitatively determined in serum by an enzyme-linked immunosorbent assay (ELISA). Individual PK parameter values were derived by non-compartmental methods using a validated PK analysis program (Kinetica™ 4.4.1 within eToolbox [version 2.6.1]).
Time Frame: Day 1 to Day 84
Population: PK evaluable Population: All participants who received at least one dose of drug and had adequate PK profiles.
Measure: Median (Full Range); unit: h
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 36 | 38
h | 2.00 [1.4 to 6.0] | 2.50 [1.4 to 6.0]

3. Secondary Outcome: Terminal Elimination Half Life (T-HALF) of Ipilimumab Manufactured by Process C Relative to the T-HALF of Ipilimumab Manufactured by Process B - Evaluable Pharmacokinetic Population
Description: The single-dose Pharmacokinetic parameters of ipilimumab were derived from serum concentration versus time data. T-HALF was measured from first dose to end of the induction period (4 doses) in day(s). Samples were obtained at 0 hour (predose) on Days 1, 2, 3, 4, and Weeks 2, 3, 4, 7, and 10; Day 1, samples were also obtained 1 h 30 minutes (min), 2 h, 2 h 30 min, 3 h 30 min, 4 h 30 min, and 6 h post dose. In calculating PK parameters, predose concentrations and concentrations prior to first quantifiable concentration below the lower limit of quantitation (LLOQ) were treated as "missing" for the calculation of summary statistics. Drug was quantitatively determined in serum by an enzyme-linked immunosorbent assay (ELISA). Individual PK parameter values were derived by non-compartmental methods using a validated PK analysis program (Kinetica™ 4.4.1 within eToolbox [version 2.6.1]).
Time Frame: Day 1 to Day 84
Population: PK evaluable Population: All participants who received at least one dose of drug and had adequate PK profiles.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 33 | 36
days | 15.45 (6.93) | 15.23 (8.73)

4. Secondary Outcome: Clearance (CLT) of Ipilimumab Manufactured by Process C Relative to the CLT of Ipilimumab Manufactured by Process B - Evaluable Pharmacokinetic Population
Description: The single-dose Pharmacokinetic parameters of ipilimumab were derived from serum concentration versus time data. CLT was measured from first dose to end of the induction period (4 doses) in milliliters per hour (mL/h). Samples were obtained at 0 hour (predose) on Days 1, 2, 3, 4, and Weeks 2, 3, 4, 7, and 10; Day 1, samples were also obtained 1 h 30 minutes (min), 2 h, 2 h 30 min, 3 h 30 min, 4 h 30 min, and 6 h post dose. In calculating PK parameters, predose concentrations and concentrations prior to first quantifiable concentration below the lower limit of quantitation (LLOQ) were treated as "missing" for the calculation of summary statistics. Drug was quantitatively determined in serum by an enzyme-linked immunosorbent assay (ELISA). Individual PK parameter values were derived by non-compartmental methods using a validated PK analysis program (Kinetica™ 4.4.1 within eToolbox [version 2.6.1]).
Time Frame: Day 1 to Day 84
Population: PK evaluable Population: All participants who received at least one dose of drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 33 | 36
mL/h | 12.590 (45) | 12.934 (53)

5. Primary Outcome: Area Under the Serum Concentration-time Curve (AUC) From Time Zero to Day 21, AUC(0-21d), of Ipilimumab Manufactured by Process C Relative to the AUC(0-21d) of Ipilimumab Manufactured by Process B - Evaluable Pharmacokinetic Population
Description: The single-dose pharmacokinetic parameters of ipilimumab were derived from serum concentration versus time data. AUC(0-21d) was measured from first dose to end of the induction period as micrograms*hours per milliliter (μg*h/mL). Samples were obtained at 0 hour (predose) on Days 1, 2, 3, 4, and Weeks 2, 3, 4, 7, and 10; Day 1, samples were also obtained 1 h 30 minutes (min), 2 h, 2 h 30 min, 3 h 30 min, 4 h 30 min, and 6 h post dose. In calculating PK parameters, predose concentrations and concentrations prior to first quantifiable concentration below the lower limit of quantitation (LLOQ) were treated as "missing" for the calculation of summary statistics. Drug was quantitatively determined in serum by an enzyme-linked immunosorbent assay (ELISA). Individual PK parameter values were derived by non-compartmental methods using a validated PK analysis program (Kinetica™ 4.4.1 within eToolbox [version 2.6.1]).
Time Frame: Day 1 to Day 84
Population: PK evaluable Population: All participants who received at least one dose of drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 33 | 36
μg*h/mL | 40374.47 (25) | 40085.9 (29)
Statistical Analysis 1: Comparison: Ipilimumab (Process B) vs Ipilimumab (Process C); Biocomparability of ipilimumab Process C to ipilimumab Process B was to be concluded if the 90% confidence intervals (CIs) for the ratio of geometric means for ipilimumab Cmax were contained within 80% to 125%. Point estimates and 90% CIs were constructed for the ratio of geometric means (Process C/Process B) for ipilimumab Cmax; Test type: Superiority or Other; Least squared linear regression; Ratio of adjusted geometric mean = 1.032, 90% CI 2-sided [0.922 to 1.156]

6. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Ipilimumab Manufactured by Process C Relative to the Vss of Ipilimumab Manufactured by Process B - Evaluable Pharmacokinetic Population
Description: The single-dose Pharmacokinetic parameters of ipilimumab were derived from serum concentration versus time data. Vss was measured from first dose to end of the induction period (4 doses) in liter(s) (L). Samples were obtained at 0 hour (predose) on Days 1, 2, 3, 4, and Weeks 2, 3, 4, 7, and 10; Day 1, samples were also obtained 1 h 30 minutes (min), 2 h, 2 h 30 min, 3 h 30 min, 4 h 30 min, and 6 h post dose. In calculating PK parameters, predose concentrations and concentrations prior to first quantifiable concentration below the lower limit of quantitation (LLOQ) were treated as "missing" for the calculation of summary statistics. Drug was quantitatively determined in serum by an enzyme-linked immunosorbent assay (ELISA). Individual PK parameter values were derived by non-compartmental methods using a validated PK analysis program (Kinetica™ 4.4.1 within eToolbox [version 2.6.1]).
Time Frame: Day 1 to Day 84
Population: PK evaluable Population: All participants who received at least one dose of drug and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 33 | 36
L | 6.06 (21) | 5.96 (32)

7. Secondary Outcome: Best Overall Tumor Response Per Investigator Based on Modified World Health Organization (mWHO) Criteria - All Randomized Participants
Description: Overall Response (OR) was determined as the combination of assessments of index and non-index lesions using mWHO criteria which were: Complete Response=complete disappearance of all lesions; Partial Response=decrease, relative to baseline, of 50% or greater in the sum of the products of the two largest perpendicular diameters of all index lesions, in the absence of Complete Response; Stable Disease=does not meet criteria for complete or partial response, in the absence of progressive disease, or a decrease or tumor stabilization of one or more non-index lesions; Progressive Disease (Progression)=at least 25% increase in the sum of the products of all index lesions (taking as reference the smallest sum recorded at or following baseline) and/or the appearance of any new lesion(s), or progression of non-index lesion(s). OR was measured across the entire study from Day 1 to the last patient, last visit (2009 to 2012)
Time Frame: Day 1 to last patient, last visit, approximately 3 years
Population: All participants randomized to a treatment arm who received at least 1 dose of ipilimumab as randomized with measurable disease at baseline, at least one baseline assessment and one on-treatment tumor assessment, no resection of index lesions.
Measure: Number; unit: participants
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 36 | 37
participants
  Complete Response mWHO | 0 | 1
  Partial Response mWHO | 4 | 10
  Stable Disease mWHO | 11 | 7
  Progression mWHO | 14 | 17
  Unable to determine mWHO | 7 | 2

8. Secondary Outcome: Best Overall Tumor Response Per Investigator Based on Immune-related (ir) Response Criteria (RC) - All Randomized Participants
Description: ir RC=modifications of mWHO criteria reflecting clinical experience with ipilimumab in over 20 completed and/or ongoing clinical studies. irRC were designed to capture clinical activity of ipilimumab immunotherapy that may not be adequately addressed by the mWHO criteria. irComplete Response (irCR): Complete disappearance of all index and non-index lesions. irPartial Response (irPR): Decrease, relative to baseline, of 50% or greater in the sum of the products of the two largest perpendicular diameters of all index and all new measurable lesions in the absence of irCR, non-index lesions not considered. irStable Disease (irSD): Does not meet criteria for irCR or irPR, in the absence of progressive disease (irPD). irProgressive Disease (irPD): At least 25% increase in Tumor Burden when compared to sum of the products of diameters of lesions at nadir.
Time Frame: Day 1 to last patient, last visit, approximately 3 years
Population: All participants randomized to a treatment arm who received at least 1 dose of ipilimumab as randomized with measurable disease at baseline, at least one baseline assessment and one on-treatment tumor assessment, no resection of index lesions, and for irRC, no resection of new lesions.
Measure: Number; unit: participants
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 33 | 34
participants
  ir Complete Response | 0 | 1
  ir Partial Response | 2 | 9
  ir Stable Disease | 11 | 8
  ir Progression | 14 | 14
  Unable to determine | 6 | 2

9. Secondary Outcome: Median Overall Survival Following First Ipilimumab Dose - All Treated Participants
Description: Overall survival (OS) was defined as the time between the first dose of study treatment and death and was analyzed using Kaplan-Meier methods, with participants who had not died censored at the last date known to be alive. Overall survival was measured in months.
Time Frame: Week 1 (first dose) to last patient, last visit, approximately 3 years
Population: All participants who received at least one dose of ipilimumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 37 | 38
months | 20.58 [8.55 to NA] — survival plateau close to 50%, therefore upper limit was not calculable | 24.79 [21.04 to 36.57]

10. Secondary Outcome: Model Estimates of Mean Absolute Lymphocyte Count at Each Nominal Ipilimumab Induction Dose and at End of the Induction Dosing Period
Description: Absolute lymphocyte counts (ALC) were obtained throughout the study as part of the hematology panel. Results collected from 28 days prior to the first infusion of ipilimumab through the end of the Induction-Dosing Period were included in the analyses of ALC. Mean ALC was estimated via an extended linear model, with linear splines and a spatial exponential within-patient correlation structure. Lymphocytes were measured as 1000 cells per micro liter (c/µL).
Time Frame: Day 0 (prior to first dose) to Day 84
Population: All participants in the Pharmacodynamic data set with: (1) a baseline ALC evaluation; and (2) at least 1 post-baseline ALC evaluation (after the date of first dose).
Measure: Mean (95% Confidence Interval); unit: 1000 c/µL
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 37 | 38
1000 c/µL
  0 days since first dose | 1.26 [0.99 to 1.53] | 1.18 [0.92 to 1.45]
  21 days since first dose | 1.67 [1.40 to 1.94] | 1.74 [1.47 to 2.00]
  42 days since first dose | 1.79 [1.51 to 2.07] | 1.86 [1.58 to 2.13]
  63 days since first dose | 2.07 [1.79 to 2.36] | 1.94 [1.66 to 2.22]
  84 days since first dose | 1.89 [1.52 to 2.27] | 2.01 [1.62 to 2.39]
Statistical Analysis 1: Comparison: Ipilimumab (Process B) vs Ipilimumab (Process C); Time-by-process interaction. Null hypothesis that the pattern of mean ALC values over time is the same for both processes; Test type: Superiority or Other; p = 0.85, F-test — Not corrected for multiple testing; numerator 5 degrees freedom, denominator 782 degrees freedom; omnibus conditional F-test = 0.40
Statistical Analysis 2: Comparison: Ipilimumab (Process B) vs Ipilimumab (Process C); Overall time effect. Null hypothesis of no mean ALC changes over time in either process group (treatment arm); Test type: Superiority or Other; p < 0.0001, F-test; numerator 10 degrees freedom, denominator 782 degrees freedom; F-statistic = 4.35

11. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and AEs Leading to Discontinuation
Description: Adverse events (AEs) and Serious AEs (SAEs) were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse events version 3.0. Medical Dictionary for Regulatory Activities (MedDRA) version 15.1 was used. Note there is a difference in number of participants with an SAE in this outcome measure and the number listed in the Adverse Events Section of this document. This is because the SAEs reported in the xml upload of the Adverse Events section includes additional participants who reported SAEs after the clinical study report database was closed.
Time Frame: Day 1 to last patient, last visit, approximately 3 years
Population: All participants who received at least 1 dose of ipilimumab.
Measure: Number; unit: participants
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 37 | 38
participants
  Participants with at least 1 AE | 37 | 38
  Participants with at least 1 treatment related AE | 33 | 36
  Participants with at least 1 SAE | 22 | 24
  Participants with at least 1 treatment related SAE | 10 | 13
  AE leading to discontinuation | 14 | 12
  Participants who died | 17 | 20

12. Secondary Outcome: Number of Participants Who Developed Antibodies and Neutralizing Antibodies
Description: Electrochemiluminescent (ECL) Immunoassay was used to detect human anti-human ipilimumab antibodies (HAHA) in serum. Blood samples were collected prior to the start of each ipilimumab infusion at Weeks 1, 4, 7, 10, 24, and at end of treatment. Those participants who were positive HAHA on treatment were then tested for presence of neutralizing antibodies.
Time Frame: Prior to start of drug Week 1 to Week 24 on treatment or end of treatment
Population: Participants who received study drug and had HAHA data prior to infusion in Week 1 and while on treatment.
Measure: Number; unit: participants
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 34 | 36
participants
  Positive HAHA on treatment | 0 | 2
  Neutralizing antibodies present | 0 | 0

13. Secondary Outcome: Mean Change From Baseline in Sitting Systolic and Diastolic Blood Pressure - All Treated Participants up to Data Cutoff
Description: Systolic and Diastolic blood pressure were measured in millimeters of mercury (mmHg) and were obtained after the participant had been seated for 5 minutes. Vital sign measurements were collected at Screening (baseline), Weeks 1, 4, 7, 10, 12, 24 and every 12 weeks thereafter in the Maintenance Phase, and at the End of Treatment visit. The change from baseline in blood pressure one hour post end of infusion at the end of induction Period, Week 36 of Maintenance Period, and end of treatment, up to data cutoff for July 2010 are presented below.
Time Frame: Screening to data cut off for July 2010, approximately 36 Weeks
Population: All participants who received at least 1 dose of ipilimumab and had available data at baseline and the specific timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 10 | 12
mmHg
  Diastolic at End of Induction (N=10, 12) | -1.6 (10.1) | -1.4 (9.7)
  Diastolic at Week 36 of Maintenance (N=7, 7) | -7.0 (14.1) | -5.6 (6.8)
  Diastolic at End of Treatment (N=6,7) | 7.5 (7.1) | 2.3 (12.4)
  Systolic at End of Induction (N=10, 12) | -4.1 (19.6) | -8.6 (21.0)
  Systolic at Week 36 of Maintenance (N=7, 7) | -5.7 (31.5) | -8.3 (18.3)
  Systolic at End of Treatment (N=6,7) | 11.5 (13.3) | -2.1 (14.7)

14. Secondary Outcome: Mean Change From Baseline in Sitting Pulse Rate - All Treated Participants up to Data Cutoff
Description: Pulse Rate was measured in beats per minute (bpm) and was obtained after the participant had been seated for 5 minutes. Vital sign measurements were collected at Screening (baseline), Weeks 1, 4, 7, 10, 12, 24 and every 12 weeks thereafter in the Maintenance Phase, and at the End of Treatment visit. The change from baseline in blood pressure one hour post end of infusion at the end of induction Period, Week 36 of Maintenance Period, and end of treatment, up to data cutoff for July 2010 are presented below.
Time Frame: Screening to data cut off for July 2010, approximately 36 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 10 | 24
bpm
  Pulse Rate at End of Induction (N=10, 24) | -4.3 (11.1) | -3.3 (11.1)
  Pulse Rate at Week 36 (N=7,7)) | -7.7 (15.3) | -7.1 (8.8)
  Pulse Rate at end of treatment (N=6,7) | 25.5 (15.8) | 12.3 (10.5)

15. Secondary Outcome: Number of Participants With 2-Grade or Greater Shift From Baseline (Worsening) in Hematology Laboratory Safety Tests - All Treated Participants
Description: Common Terminology Criteria (CTC), Version 3 used to assess parameters. Lower limit of normal (LLN); grams per deciliter (g/dL); Grade (GR); cells per microliter (c/µL). Hemoglobin Gr 1:<LLN to 10.0 g/dL, Gr 2:<10.0 to 8.0 g/dL, Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL. Absolute neutrophil (ANC) and ANC plus bands: Gr 1:<LLN to 1.5*10^3 c/µL, Gr 2:<1.5 to 1.0*10^3 c/µL, Gr 3:<1.0 to 0.5*10^3 c/µL, Gr 4:<0.5*10^3 c/µL. Platelet count Gr 1:LLN to 75.0*10^9 c/L, Gr 2:<75.0 to 50.0*10^9 c/L, Gr 3:<50.0 to 25.0*10^9 c/L, Gr 4:<25.0 to 10^9 c/L. Lymphocytes Gr 1: <1.5 to 0.8 *10^3 c/µL, Gr 2 <0.8 to 0.5 *10^3 c/µL, Gr 3: <0.5 to 0.2 *10^3 c/µL, Gr 4: <0.2*10^3 c/µL. Leukocytes Gr 1:<LLN to 3.0 *10^3 c/µL, Gr 2; <3.0 to 2.0 *10^3 c/µL, Gr 3: <2.0 to 1.0 *10^3 c/µL, Gr 4: <1.0 *10^3 c/µL. Baseline is screening or Day 1, prior to dosing.
Time Frame: Screening to data cut off for July 2010, approximately 36 Weeks
Population: All participants who received at least 1 dose of ipilimumab and had available data at baseline and post baseline.
Measure: Number; unit: participants
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 37 | 38
participants
  Hemoglobin (N=37, 38) | 2 | 3
  Lymphocytes (N=37, 38) | 3 | 3
  Neutrophils, Absolute (N=31, 36) | 0 | 2
  Neutrophils + bands, Absolute (N=31, 36) | 0 | 1
  Platelet Count (N=37, 38) | 0 | 1

16. Secondary Outcome: Number of Participants With 2-Grade or Greater Shift From Baseline (Worsening) in Chemistry Laboratory Safety Tests (Non-electrolyte) - All Treated Participants
Description: Alanine transaminase (ALT); Aspartate aminotransferase (AST); Alkaline phosphatase (ALP); upper limits of normal (ULN). ALT Gr 1:>1.0 to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. AST Gr 1: >1.0 to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. Total bilirubin Gr 1: >1.0 to 1.5*ULN; Gr 2: >1.5 to 3.0*ULN; Gr 3: >3.0 to 10..0*ULN; Gr 4: >10.0.0*ULN. ALP (U/L) Gr1:>1.0 to 2.5*ULN, Gr2:>2.5 to 5.0*ULN, Gr3:>5.0 to 20.0*ULN, Gr4:>20.0*ULN. Albumin (low) Gr 1:<LLN to 3 g/dL; Gr 2: <3.0 - 2.0 g/L; Gr 3: < 2 g/dL. Creatinine Gr 1: >1 - 1.5*ULN; Gr 2: >1.5 - 3.0*ULN; Gr 3: >3.0- 6.0*ULN; Gr 4: >6.0*ULN. Lipase (U/L) Gr 1: 1.0 to 1.5*ULN; Gr 2: >1.5 to 2.0*ULN; Gr 3: 2.0 to 5; Gr 4: >5*ULN. Amylase (U/L) Gr 1: >ULN to 1.5*ULN; Grade 2 >1.5 to 2.0*ULN, Grade 3 >2.0 to 5.0*ULN, Grade 4 >5.0*ULN. Baseline was screening or Day 1, prior to first dose of drug.
Time Frame: Screening to data cut off for July 2010, approximately 36 Weeks
Population: All participants who received at least 1 dose of ipilimumab and had available data at baseline and post baseline.
Measure: Number; unit: participants
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 37 | 38
participants
  ALT (N=36, 37) | 2 | 1
  AST (N=36, 37) | 2 | 1
  Alkaline Phosphatase (N=36, 37) | 2 | 1
  Amylase (N=35, 35) | 0 | 2
  Lipase (N=10, 14) | 0 | 1
  Albumin (N=36, 37) | 7 | 8
  Creatinine (N= 37, 37) | 2 | 1
  Bilirubin (N=36, 37) | 2 | 0

17. Secondary Outcome: Number of Participants With 2-Grade or Greater Shift From Baseline (Worsening) in Electrolyte Laboratory Safety Tests - All Treated Participants
Description: Sodium high (H) Gr 1:>ULN - 150; Gr 2: >150 - 155; Gr 3: >155 - 160; Gr 4: >160 mmol/L; Sodium low(L) Gr 1:<LLN - 130; Gr 3: <130 - 120; Gr 4: <120 mmol/L. Potassium (H) Gr 1: >ULN - 5.5; Gr 2: >5.5 - 6.0; Gr 3: > 6.0 - 7.0; Gr 4: >7.0 mmol/L; Potassium (L) Gr 1: <LLN - 3.0; Gr 2: <LLN - 3.0; Gr 3: < 3.0 - 2.5; Gr 4: <2.5 mmol/L. Bicarbonate Gr1: 16-<LLN, Gr2: 11-16, Gr3, 8-11, Gr4: <8 milliequivalents per liter (mEq/L). Phosphorus Gr 1: 2.5 - <LLN, Gr2 2.0-<2.5, Gr3: 1.0-<2.0, Gr4: <1.0. Calcium (L) Gr 1: <LLN to 8.0; Gr2: 7.0 - 8.0; Gr3: 6.0-7.0; Gr 4: <6.0 mg/dL; calcium (H) Gr1:>ULN - 11.5, Gr2:>11.5 - 12.5, Gr3: 12.5 - 13.5, Gr4: >13.5. Baseline is screening or Day 1, prior to first dose of drug.
Time Frame: Screening to data cut off for July 2010, approximately 36 Weeks
Population: All participants who received at least 1 dose of ipilimumab and had available data at baseline and post baseline.
Measure: Number; unit: participants
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Number analyzed (Participants) | 37 | 38
participants
  Sodium (low) (N=37, 37) | 4 | 6
  Potassium (low) (N=36, 37) | 1 | 2
  Potassium (high) (N=36, 37) | 0 | 1
  Calcium (low) (N=37, 37) | 1 | 7
  Inorganic Phosphorus (N=37,37) | 9 | 7
  Bicarbonate (N=37, 37) | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to last patient, last visit, approximately 3 years.
Description: SAEs and AEs 5% threshold up to last patient, last visit (31 Oct 2012) were in primary endpoint posting. Therefore, SAEs and AEs have not changed with this current PRS update from Maintenance Period. SAE/AE upload includes SAEs reported after the data cut off for the clinical study report and thus differs slightly from data in Outcome measure 11.
Arm/Group | Ipilimumab (Process B) | Ipilimumab (Process C)
Serious Adverse Events (participants affected / at risk) | 24/37 | 26/38
Other Adverse Events (participants affected / at risk) | 37/37 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (Process B) (N=37) | Ipilimumab (Process C) (N=38)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Hypopituitarism (Endocrine disorders) | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Localised oedema (General disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Pyrexia (General disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Skin cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Asthenia (General disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 1
Colitis (Gastrointestinal disorders) | 4 | 8
Confusional state (Psychiatric disorders) | 2 | 1
Platelet count decreased (Investigations) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 2
Temporal arteritis (Vascular disorders) | 1 | 0
Amylase increased (Investigations) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 6
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (Process B) (N=37) | Ipilimumab (Process C) (N=38)
Abdominal distension (Gastrointestinal disorders) | 3 | 3
Blastocystis infection (Infections and infestations) | 0 | 2
Chest pain (General disorders) | 2 | 1
Chills (General disorders) | 2 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Hypoaesthesia (Nervous system disorders) | 1 | 2
Hypophysitis (Endocrine disorders) | 2 | 1
Hypotension (Vascular disorders) | 3 | 0
Influenza like illness (General disorders) | 1 | 3
Mucosal inflammation (General disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2
Syncope (Nervous system disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 7 | 13
White blood cell count decreased (Investigations) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Candidiasis (Infections and infestations) | 2 | 3
Depression (Psychiatric disorders) | 2 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Oral herpes (Infections and infestations) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Alanine aminotransferase increased (Investigations) | 6 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 5
Dizziness (Nervous system disorders) | 4 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 29 | 22
Haemoglobin decreased (Investigations) | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Oedema peripheral (General disorders) | 3 | 7
Pain (General disorders) | 6 | 4
Urinary retention (Renal and urinary disorders) | 2 | 0
Uveitis (Eye disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 12
Agitation (Psychiatric disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Dysgeusia (Nervous system disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 4 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 5 | 1
Nausea (Gastrointestinal disorders) | 14 | 19
Neutrophil count decreased (Investigations) | 1 | 2
Pyrexia (General disorders) | 7 | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 | 0
Rhinitis (Infections and infestations) | 0 | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 7
Asthenia (General disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 14 | 14
Dyspepsia (Gastrointestinal disorders) | 1 | 7
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Headache (Nervous system disorders) | 9 | 14
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hot flush (Vascular disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3
Hypothyroidism (Endocrine disorders) | 4 | 5
Mood swings (Psychiatric disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 5
Oedema (General disorders) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 5
Blood creatinine increased (Investigations) | 2 | 0
Blood testosterone decreased (Investigations) | 2 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cellulitis (Infections and infestations) | 2 | 0
Colitis (Gastrointestinal disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 3 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Flushing (Vascular disorders) | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Influenza (Infections and infestations) | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 3
Platelet count decreased (Investigations) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 24
Stomatitis (Gastrointestinal disorders) | 0 | 2
Weight increased (Investigations) | 0 | 2
Amylase increased (Investigations) | 4 | 2
Ascites (Gastrointestinal disorders) | 1 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 3
Blood bilirubin increased (Investigations) | 2 | 1
Constipation (Gastrointestinal disorders) | 9 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 7 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 21 | 25
Sinusitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 4
Urinary tract infection (Infections and infestations) | 3 | 2
Anxiety (Psychiatric disorders) | 4 | 4
Conjunctivitis (Eye disorders) | 0 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 18 | 26
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 4
Lipase increased (Investigations) | 4 | 2
Nodule (General disorders) | 2 | 3
Oral candidiasis (Infections and infestations) | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Vision blurred (Eye disorders) | 1 | 4
Weight decreased (Investigations) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.